CLINICAL TRIAL: NCT06418776
Title: A Prospective Multicenter Randomized Clinical Trial on the Treatment of Patients With Refractory or Early Relapses of Acute Myeloid Leukemia
Brief Title: IMPACT-AML: Randomized Pragmatic Clinical Trial for Relapsed or Refractory AML
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Research Center for Hematology, Russia (Network)
Collaborators: St. Petersburg State Pavlov Medical University (Other); Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Responsible Party: Principal Investigator, Elena N.Parovichnikova, General director of National Medical Research Center for Hematology, National Research Center for Hematology, Russia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMPACT-AML
Record Dates: First submitted 2024-04-09; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Refractory Acute Myeloid Leukemia; Early Relapses of Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; Relapse of AML; Refractory AML; Allogeneic Stem Cell Transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: Patients who could potentially undergo courses of intensive chemotherapy ("fit") are randomisedrandomized into two arms:
  * Arm 1 - intensive chemotherapy courses (MEC, FLAG, FLAG-Ida, FLAG-Mito)
  * Arm 2 - low intensity therapy (Aza/Dac/LDARA-C + Ven) Randomization determines the intensity of the program, but not the specific therapeutic regimen. The treatment regimen is selected by the investigators based on accepted clinical practice, the availability of appropriate drugs at the participating centers, etc., after randomization. If a patient has FLT3 gene mutations, one of the available kinase inhibitors must be added to therapy: midostaurin, gilteritinib, sorafenib.
  If remission of the AML has been achieved, patients in both groups undergo alloHSCT as soon as possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intensive arm (Active Comparator): Fit patients who could potentially undergo courses of intensive chemotherapy and are randomized to intensive chemotherapy courses
  Interventions: Other: Intensive therapy
- Low-intensive arm (Active Comparator): Fit patients who could potentially undergo courses of intensive chemotherapy and are randomized to low intensity courses
  Interventions: Other: Low intensity therapy

INTERVENTIONS:
Other: Intensive therapy — Intensive chemotherapy courses (MEC, FLAG, FLAG-Ida, FLAG-Mito)
  Arms: Intensive arm
Other: Low intensity therapy — Low intensity therapy (Aza+Ven, Dac+Ven, LDARA-C+Ven)
  Arms: Low-intensive arm

SUMMARY:
The primary objective is to evaluate the efficacy and toxicity of high versus low intensity therapy options in patients with refractory forms and early relapses of acute myeloid leukemia (R/R AML) who are scheduled for allogeneic hematopoietic stem cell transplantation (alloHSCT).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Primary refractory AML;
* Early relapsed AML;
* A signed informed consent to participate in the study.

Exclusion Criteria:

* Late relapsed AML;
* Isolated extramedullary relapse;
* MRD relapse without development of bone marrow relapse of AML;
* Acute promyelocytic leukemia;
* Previous refractoriness or loss of response during ongoing venetoclax therapy;
* Previous alloHSCT;
* Pregnancy and/or lactation period;
* Refusal of patients with preserved reproductive potential to use highly effective methods of contraception during the period of participation in the study;
* Lack of signed informed consent to participate in the study;
* Failure of the subject to follow the study protocol;
* Participation in any other clinical trial;
* Uncontrolled infectious complications;
* ECOG ≥ 3;
* History of other malignancies within the past 3 years, excluding squamous cell and basal cell skin cancers, carcinoma in situ of the cervix, breast, or other non-invasive malignancies, which, in the opinion of the investigator, are considered adequately treated and have a minimal risk of recurrence within 3 years;
* Chronic kidney disease with GFR ≤ 30 ml/min/1.73 m2 (according to the CKD-EPI Creatinine Equation);
* Severe cardiac pathology:

  1. uncontrolled arterial hypertension;
  2. stable angina III-IV functional classes;
  3. unstable angina and/or myocardial infarction less than 6 months before inclusion in the study;
  4. heart failure stages IIb-III, NYHA functional classes III-IV
  5. uncontrolled cardiac rhythm disturbances (≥ 2 grade CTCAE 5.0) or clinically significant ECG abnormalities.
* Cirrhosis classes B-C according to the Child-Pugh classification
* Increased liver function tests above the following values:

  1. Total bilirubin > 1,5 above the normal range;
  2. AST, ALT > 10 above the normal range.
* Major surgical interventions underwent less than 14 days before inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Event-free survival of patients with R/R AML depending on the use of high or low intensity therapy exposure before alloHSCT | 2 years
  Evaluation method: Kaplan-Meier curves and log-rank test, censored for transplantation

SECONDARY OUTCOMES:
Probability of achieving CR in patients with R/R AML, depending on the use of high or low intensity treatment regimens | 3 months
  Assessment method: Chi-square test
Probability of achieving a response (CR, CR with incomplete hematological recovery, morphologic leukemia- free state, partial remission) in patients with R/R AML, depending on the use of high or low intensity treatment regimens | 3 months
  Assessment method: Chi-square test
Cumulative incidence of alloHSCT in patients with R/R AML, depending on the use of high or low intensity treatment regimens | 2 years
  Evaluation method: cumulative frequency curves and Gray's test
Toxicity of high versus low intensity regimens | 3 months
  Evaluation method: Chi-square test, parametric/nonparametric tests for means
  Variables to be evaluated:
  1. Maximum degree and duration of neutropenia and/or thrombocytopenia;
  2. Development of uncontrolled/life-threatening infectious complications;
  3. Development of life-threatening hemorrhagic complications;
  4. Development of severe organ failure.
OS over the entire duration of the study, including follow-up after alloHSCT | 2 years
  Evaluation method: Kaplan-Meier curves and log-rank test
RFS in patients with R/R AML when achieving remission before alloHSCT, depending on the use of high or low intensity treatment regimens | 2 years
  Evaluation method: Kaplan-Meier curves and log-rank test
Relapse incidence in patients with R/R AML when achieving remission before performing alloHSCT, depending on the use of high or low intensity treatment regimens | 2 years
  Evaluation method: cumulative frequency curves and Gray's test
EFS of patients with R/R AML depending on the use of high or low intensity regimens, regardless of alloHSCT | 2 years
  Evaluation method: Farington-Manning test, not censored for transplantation
Statistics on discontinued participation in the protocol and premature withdrawal from the study | 2 years
  Assessment method: Chi-square test

CONTACTS AND LOCATIONS:
Locations (1):
- National Research Center for Hematology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
Each center participating in the study includes patients and fills CRF forms separately.